CLINICAL TRIAL: NCT04009590
Title: Quit4Health: Expanding the Reach of an Innovative Tobacco Control Program for Young Adults
Brief Title: Quit4Health Intervention in Supporting Smoking Cessation and Preventing Smoking Initiation in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0186; NCI-2018-03518 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0186 (Other: M D Anderson Cancer Center); R42DA035012 (NIH)
Record Dates: First submitted 2019-02-19; First posted 2019-07-05 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Cigarette Smoking; Current Smoker
MeSH Terms: conditions — Cigarette Smoking | interventions — Early Intervention, Educational; Educational Status; Methods; Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP I (Quit4Health) (Experimental): Participants utilize Quit4Health intervention that includes interactive features, coping strategies and games related to cigarettes and other tobacco products for 1 month.
  Interventions: Other: Questionnaire Administration; Behavioral: Smoking Cessation Intervention
- Group II (educational booklet) (Active Comparator): Participants read an educational booklet about cigarettes and other tobacco products for 1 month.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Read educational booklet
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group II (educational booklet)
Other: Questionnaire Administration — Ancillary studies
Behavioral: Smoking Cessation Intervention — Utilize Quit4Health
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: GROUP I (Quit4Health)

SUMMARY:
This trial studies how well Quit4Health intervention works in supporting smoking cessation and preventing smoking initiation in young adults. Quit4Health intervention may help young adults learn more about the risks of tobacco use and may help them to quit smoking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether smokers randomized to Quit4Health are more likely to quit smoking and remain tobacco-free at 6 months than subjects randomized to the education only control group.

II. To evaluate whether non-smokers who are randomized to Quit4Health are less likely to initiate tobacco usage and remain tobacco-free at 6 months than non-smokers randomized to the education only control group.

SECONDARY OBJECTIVES:

I. To evaluate whether well-established predictors of susceptibility and barriers to cessation (e.g. self-efficacy, knowledge about associated risks, normative beliefs, attitudes, resistance skills, peer pressure) and recently identified predictors of tobacco use (e.g., depression, nicotine dependence, alcohol use, risk-taking propensity) will mediate the effect of the intervention on both onset (for non-smokers) and cessation (for smokers) of tobacco use.

II. To evaluate whether, at the end-of-treatment (EOT) assessment, participants (both smokers and non-smokers) in Quit4Health will report a significantly better perception of Quit4Health (message relevance, tailoring to specific needs based on tobacco use status, motivation to quit, etc.) compared with their counterparts in the education only control arm.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants utilize Quit4Health intervention that includes interactive features, coping strategies and games related to cigarettes and other tobacco products for 1 month.

GROUP II: Participants read an educational booklet about cigarettes and other tobacco products for 1 month.

After completion of study, participants are followed at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in at least one class at Houston Community College (HCC) Central campus, West Loop campus or Spring Branch campus (cessation and prevention/advocacy groups)
* Speak and read English (cessation and prevention/advocacy groups)
* Own an Android or iOS smartphone (cessation and prevention/advocacy groups)
* Provide current and relevant contact information (cessation and prevention/advocacy groups)
* Smoked at least one cigarette (or more) in the past 30 days (cessation group)
* Have data and wifi capabilities on their mobile device (cessation and prevention/advocacy groups)
* Evidence of smoking susceptibility as defined by the Smoking Susceptibility Scale (prevention/advocacy groups)

Exclusion Criteria:

* People who score 16 or above on the Center for Epidemiologic Studies Depression (CESD) thus showing evidence of major depressive disorder (cessation and prevention/advocacy groups)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 579 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Abstinence from tobacco | At 6 months
  Any abstinence is defined as "subjective reports of abstinence from tobacco for at least 24 hours or more in the past 30 days", the 7-day point prevalence of abstinence at follow-ups will be verified by measurement of saliva cotinine. The primary analysis will compare the abstinence rates at 6 months in the control and treatment group using a 2-sample test of proportion for all smokers. A secondary analysis will involve a simple post-test analysis among smokers using logistic regression.
Susceptibility to tobacco initiation | At 6 months
  Will assess susceptibility to smoking using the measure proposed by Pierce and colleagues. Will employ similar analytic methods as in primary objective 1 to evaluate the prevalence of susceptibility at the 6-month follow-up in subjects randomized to the experimental intervention condition with respect to subjects assigned to the control condition.

SECONDARY OUTCOMES:
Mediation effect of predictors of smoking and recently identified predictors of tobacco use | Up to 6 months
  The mediation effect estimate will be computed as the product of the effect of the treatment on the mediators and the mediators on the outcome controlling for the treatment. The Bayesian mediation analysis method detailed by Yuan and MacKinnon will be used to estimate and make inference on the mediation effect.
Behavior modification | Up to 6 months
  Will evaluate the motivational appeal, educational relevance and knowledge acquired in specific modules of the app that lead to behavior modification. Similar assessments will be done among participants in the control condition with educational materials.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Prokhorov, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org